CLINICAL TRIAL: NCT04245540
Title: A Single Arm, Open-label Pilot Trial Examining the Effects of Pau d' Arco on Primary Dysmenorrhea in Reproductive Age Women
Brief Title: Effects of Pau d' Arco in Primary Dysmenorrhea
Acronym: EPAPD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RB11617
Record Dates: First submitted 2018-05-16; First posted 2020-01-29 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; dysmenorrhea; tabebuia avellanedae; tabebuia impetiginosa; pau d' arco; taheebo bark; menstrual pain; pelvic pain; menstrual cramps; painful menstruation; menstrual distress; herbal medicine; phytomedicine; complementary therapy; complementary medicine; alternative therapy; alternative medicine; traditional medicine; plant extracts; supplement
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Single arm, open-label trial evaluating safety and tolerability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): 1,050 mg per day of encapsulated Pau d' Arco taken orally for 2 months.
  Interventions: Dietary Supplement: Pau d' Arco

INTERVENTIONS:
Dietary Supplement: Pau d' Arco — Encapsulated herbal Pau d' Arco.

SUMMARY:
A single arm, open-label trial evaluating safety and tolerability of encapsulated Tabebuia avellanedae in 12 generally healthy women aged 18-45 with primary dysmenorrhea (PDM). This will be the first study evaluating the safety and tolerability of Tabebuia avellanedae in PDM. We also aim to collect proof-of-concept mechanistic data supporting the hypothesis that Tabebuia avellanedae reduces PGE2 concentration in vivo in women with PDM.

DETAILED DESCRIPTION:
This is a single arm, open-label trial evaluating safety and tolerability of 1,050 mg/day of encapsulated Tabebuia avellanedae every day for 2 months, as well as effects of the treatment on quality of life, pain intensity, and pain interference, in 12 generally healthy women aged 18-45 with PDM. Outcomes of this study include questionnaires to evaluate: safety and tolerability using standardized adverse events scales (primary); participant reported measurements of quality of life, pain intensity, and pain interference around menses collected on validated instruments (secondary); and blood concentration of PGE2 and high-sensitivity C-reactive protein (tertiary). The protocol followed the SPIRIT guidelines and fulfilled the SPIRIT checklist.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* Ages 18-45
* Presence of primary dysmenorrhea
* Has a 'smart' phone and is willing to download and use an electronic application for use during the study.
* Willing to take a non-hormonal form of birth control throughout the trial period (abstinence, condom, diaphragm, or copper IUD (ParaGard))
* Lives in the Portland area
* Able to speak, read and write English
* Has reliable transportation to clinic
* Willing to have four fasting blood draws taken
* Wiling to collect menstrual fluid in a Diva© cup on the first day of menstruation and ability to deliver it to the clinic on the same day
* Ability to receive and complete electronic VAS scales
* Pain scale rating of 6 or higher on the VAS scale
* Monthly pain that correlates with menstruation

Exclusion Criteria:

* Presence of secondary dysmenorrhea
* General health measures outside of normal range:

  * Blood pressure readings obtained at the Screening Visit reveal hypotension (≤90/60 mmHg) or hypertension (≥140/90 mmHg).
  * Aspartate aminotransferase (AST) < 8 U/L or > 48 U/L at the Screening Visit.
  * Alanine aminotransferase (AST) < 7 U/L or > 55 U/L at the Screening Visit.
  * Estimated glomerular filtration rate (eGFR) < 90 ml/min/1.73m2 at the Screening Visit.
  * An INR value > 1.1 at the Screening Visit.
  * A red blood cell count < 3.90 million cells/mcL or > 5.03 million cells/mcL.
  * A hemoglobin value of < 12 g/dL (120 g/L) or > 15.5 g/dL (155 g/L).
  * A hematocrit value of < 34.9% or > 44.5%.
  * A white blood cell count < 3.5 billion cells/L (3,500 cells/mcL) or > 10.5 billion cells/L (10,500 cells/mcL)
  * A platelet count < 150 billion/L (150,000/mcL) or > 450 billion/L (450,000 mcL).
* Women who are nursing, pregnant, or planning pregnancy in the next four months
* Difficulty swallowing or aversion to capsules, tablets, or pills
* Currently taking, and unwilling to discontinue, NSAIDs (Aspirin, Ibuprofen)
* Currently taking dietary supplements with any of the following ingredients in amounts over 250 mg/day: cinnamon, garlic, ginger, turmeric, and/or curcumin
* Consumption of >1 alcoholic drink per day, during the study period
* Currently taking any anticoagulation medications (Warfarin/Coumadin)
* Currently taking, or have taken in the past two months, hormonal forms of birth control
* Unwillingness, or inability, to take a monthly pregnancy test during the timeline of the study (3 pregnancy tests)
* Past or present medical history of any of the following:

  * Blood clotting disorders (von Willebrand disease, Hemophilia A, Hemophilia B, etc.)
  * Liver disease (cirrhosis, hepatitis, liver failure, jaundice, liver cancer, etc.)
  * Kidney disease (chronic kidney disease, polycystic kidney disease, etc.)
  * Cardiac disease (hypertension, heart failure, cardiomyopathy, etc.)
  * Anemia (iron deficiency, sickle cell, aplastic, etc.)
  * Inflammatory bowel disease
  * Irritable bowel syndrome
  * Endometriosis
  * Obstructive endometrial polyps
  * Chronic pelvic inflammatory disease
  * Polycystic Ovarian Syndrome
  * Adenomyosis
  * Intrauterine or pelvic adhesions
  * Congenital obstructive mullerian malformations
  * Cervical stenosis
  * Use of an intrauterine contraceptive device that causes pain
  * Pelvic congestion syndrome
  * Reproductive cancer (uterine cancer, ovarian cancer, endometrial cancer, etc.)
  * Ovarian cysts
  * Fibroids
  * Uteropelvic junction obstruction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must have the ability to menstruate to participate in the current study.
Enrollment: 12 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Red Blood Cell Count | Mean change in Screening RBC count to 4 weeks.
  Red blood cell count will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 3.80-5.10 Million/uL. Red blood cell (RBC) count of less than 3.80 Million/uL will be considered as new onset anemia and will result in the participant being withdrawn from the study. This measure will be reported as: "Number of participants with normal RBC count levels," "Number of participants with abnormal RBC count values," and "Number of participants withdrawn from the study based on decreased RBC count values."
Red Blood Cell Count | Mean change in Screening RBC count to 8 weeks.
  Red blood cell count will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 3.80-5.10 Million/uL. Red blood cell (RBC) count of less than 3.80 Million/uL will be considered as new onset anemia and will result in the participant being withdrawn from the study. This measure will be reported as: "Number of participants with normal RBC count levels," "Number of participants with abnormal RBC count values," and "Number of participants withdrawn from the study based on decreased RBC count values."
Red Blood Cell Count | Mean change in 4 weeks RBC count to 8 weeks.
  Red blood cell count will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 3.80-5.10 Million/uL. Red blood cell (RBC) count of less than 3.80 Million/uL will be considered as new onset anemia and will result in the participant being withdrawn from the study. This measure will be reported as: "Number of participants with normal RBC count levels," "Number of participants with abnormal RBC count values," and "Number of participants withdrawn from the study based on decreased RBC count values."
Hemoglobin | Mean change in Screening Hemoglobin g/dL to 4 weeks.
  Hemoglobin is a protein in red blood cells that carries oxygen throughout the body. Hemoglobin will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 11.7-15.5 grams per deciliter (g/dL). Hemoglobin of less than 11.7 g/dL or greater than 15.5 g/dL will be considered as abnormal. This measure will be reported as: "Number of participants with normal Hemoglobin levels" and "Number of participants with abnormal Hemoglobin values."
Hemoglobin | Mean change in Screening Hemoglobin g/dL to 8 weeks.
  Hemoglobin is a protein in red blood cells that carries oxygen throughout the body. Hemoglobin will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 11.7-15.5 grams per deciliter (g/dL). Hemoglobin of less than 11.7 g/dL or greater than 15.5 g/dL will be considered as abnormal. This measure will be reported as: "Number of participants with normal Hemoglobin levels" and "Number of participants with abnormal Hemoglobin values."
Hemoglobin | Mean change in 4 weeks Hemoglobin g/dL to 8 weeks.
  Hemoglobin is a protein in red blood cells that carries oxygen throughout the body. Hemoglobin will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 11.7-15.5 grams per deciliter (g/dL. Hemoglobin of less than 11.7 g/dL or greater than 15.5 g/dL will be considered as abnormal. This measure will be reported as: "Number of participants with normal Hemoglobin levels" and "Number of participants with abnormal Hemoglobin values."
Hematocrit | Mean change in Screening Hematocrit % to 4 weeks.
  Hematocrit is the ratio of the volume of red blood cells to the total volume of blood. Hematocrit will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 35.0-45.0 %. Hemoglobin of less than 35.0% or greater than 45.0% will be considered as abnormal. This measure will be reported as: "Number of participants with normal Hemotocrit % levels" and "Number of participants with abnormal Hematocrit % values."
Hematocrit | Mean change in Screening Hematocrit % to 8 weeks.
  Hematocrit is the ratio of the volume of red blood cells to the total volume of blood. Hematocrit will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 35.0-45.0 %. Hemoglobin of less than 35.0% or greater than 45.0% will be considered as abnormal. This measure will be reported as: "Number of participants with normal Hemotocrit % levels" and "Number of participants with abnormal Hematocrit % values."
Hematocrit | Mean change in 4 weeks Hematocrit % to 8 weeks.
  Hematocrit is the ratio of the volume of red blood cells to the total volume of blood. Hematocrit will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 35.0-45.0 %. Hemoglobin of less than 35.0% or greater than 45.0% will be considered as abnormal. This measure will be reported as: "Number of participants with normal Hemotocrit % levels" and "Number of participants with abnormal Hematocrit % values."
Mean Corpuscular Volume | Mean change in Screening MCV fL to 4 weeks.
  Mean Corpuscular Volume (MCV) measures the average red blood cell volume. MCV will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 80.0-100.0 femtolitre (fL). MCV of less than 80.0 fL or greater than 100.0 fL will be considered as abnormal. This measure will be reported as: "Number of participants with normal MCV fL levels" and "Number of participants with abnormal MCV fL values."
Mean Corpuscular Volume | Mean change in Screening MCV fL to 8 weeks.
  Mean Corpuscular Volume (MCV) measures the average red blood cell volume. MCV will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 80.0-100.0 femtolitre (fL). MCV of less than 80.0 fL or greater than 100.0 fL will be considered as abnormal. This measure will be reported as: "Number of participants with normal MCV fL levels" and "Number of participants with abnormal MCV fL values."
Mean Corpuscular Volume | Mean change in 4 weeks MCV fL to 8 weeks.
  Mean Corpuscular Volume (MCV) measures the average red blood cell volume. MCV will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 80.0-100.0 femtolitre (fL). MCV of less than 80.0 fL or greater than 100.0 fL will be considered as abnormal. This measure will be reported as: "Number of participants with normal MCV fL levels" and "Number of participants with abnormal MCV fL values."
Mean Corpuscular Hemoglobin | Mean change in Screening MCH pg to 4 weeks.
  Mean Corpuscular Hemoglobin (MCH) measures the average mass of hemoglobin per red blood cell. MCH will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 27.0-33.0 picogram (pg). MCH of less than 27.0 pg or greater than 33.0 pg will be considered as abnormal. This measure will be reported as: "Number of participants with normal MCH pg levels" and "Number of participants with abnormal MCH pg values."
Mean Corpuscular Hemoglobin | Mean change in Screening MCH pg to 8 weeks.
  Mean Corpuscular Hemoglobin (MCH) measures the average mass of hemoglobin per red blood cell. MCH will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 27.0-33.0 picogram (pg). MCH of less than 27.0 pg or greater than 33.0 pg will be considered as abnormal. This measure will be reported as: "Number of participants with normal MCH pg levels" and "Number of participants with abnormal MCH pg values."
Mean Corpuscular Hemoglobin | Mean change in 4 weeks MCH pg to 8 weeks.
  Mean Corpuscular Hemoglobin (MCH) measures the average mass of hemoglobin per red blood cell. MCH will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 27.0-33.0 picogram (pg). MCH of less than 27.0 pg or greater than 33.0 pg will be considered as abnormal. This measure will be reported as: "Number of participants with normal MCH pg levels" and "Number of participants with abnormal MCH pg values."
Mean Corpuscular Hemoglobin Concentration | Mean change in 4 weeks MCH pg to 8 weeks.
  Mean Corpuscular Hemoglobin Concentration (MCHC) measures the average mass of hemoglobin per red blood cell. MCH will be collected through a Complete Blood Count (CBC) test. Normal ranges for this test are 27.0-33.0 picogram (pg). MCH of less than 27.0 pg or greater than 33.0 pg will be considered as abnormal. This measure will be reported as: "Number of participants with normal MCH pg levels" and "Number of participants with abnormal MCH pg values."
Recruitment and retention. | Percent change from Baseline Recruitment to 8 weeks.
  Recruitment of 12 women with primary dysmenorrhea and retention of at least 10 participants throughout the course of the study. Reported as number of recruited participants, number of excluded participants, and number of drop out participants.
Incidence of Intervention-attributable Adverse Events | Percent change from Baseline Intervention-attributable Adverse Events to 4 weeks.
  Self-reported adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events. Reported as: New onset "FDA serious" adverse events; New onset "moderate" adverse events; all reported adverse events
Incidence of Intervention-attributable Adverse Events | Percent change from Baseline Intervention-attributable Adverse Events to 8 weeks.
  Self-reported adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events. Reported as: New onset "FDA serious" adverse events; New onset "moderate" adverse events; all reported adverse events
Incidence of Intervention-attributable Adverse Events | Percent from 4 weeks Intervention-attributable Adverse Events to 8 weeks.
  Self-reported adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events. Reported as: New onset "FDA serious" adverse events; New onset "moderate" adverse events; all reported adverse events
Aspartate aminotransferase (AST) | Mean change in Screening AST values at 4 weeks.
  Aspartate aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. This value is reported as cubic rack units (U) per liter (L); (U/L). Normal ranges are 10-30 U/L. Any participant with a value of 2 times or higher of the upper end of this range (60 U/L or greater) will be withdrawn from the study per study stopping criteria. This value will be reported as: "Number of participants with normal AST levels," "Number of participants with abnormal AST values," and "Number of participants withdrawn from the study based on elevated AST values."
Aspartate aminotransferase (AST) | Mean change in Screening AST values at 8 weeks.
  Aspartate aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. This value is reported as cubic rack units (U) per liter (L); (U/L). Normal ranges are 10-30 U/L. Any participant with a value of 2 times or higher of the upper end of this range (60 U/L or greater) will be withdrawn from the study per study stopping criteria. This value will be reported as: "Number of participants with normal AST levels," "Number of participants with abnormal AST values," and "Number of participants withdrawn from the study based on elevated AST values."
Aspartate aminotransferase (AST) | Mean change in 4 weeks AST values at 8 weeks.
  Aspartate aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. This value is reported as cubic rack units (U) per liter (L); (U/L). Normal ranges are 10-30 U/L. Any participant with a value of 2 times or higher of the upper end of this range (60 U/L or greater) will be withdrawn from the study per study stopping criteria. This value will be reported as: "Number of participants with normal AST levels," "Number of participants with abnormal AST values," and "Number of participants withdrawn from the study based on elevated AST values."
Alanine aminotransferase (ALT) | Mean change in Screening ALT values at 4 weeks.
  Alanine aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. This value is reported as cubic rack units (U) per liter (L); (U/L). Normal ranges are 6-29 U/L. Any participant with a value of 2 times or higher of the upper end of this range (58 U/L or greater) will be withdrawn from the study per study stopping criteria. This value will be reported as: "Number of participants with normal ALT levels," "Number of participants with abnormal ALT values," and "Number of participants withdrawn from the study based on elevated ALT values."
Alanine aminotransferase (ALT) | Mean change in Screening ALT values at 8 weeks.
  Alanine aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. This value is reported as cubic rack units (U) per liter (L); (U/L). Normal ranges are 6-29 U/L. Any participant with a value of 2 times or higher of the upper end of this range (58 U/L or greater) will be withdrawn from the study per study stopping criteria. This value will be reported as: "Number of participants with normal ALT levels," "Number of participants with abnormal ALT values," and "Number of participants withdrawn from the study based on elevated ALT values."
Alanine aminotransferase (ALT) | Mean change in 4 weeks ALT values at 8 weeks.
  Alanine aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. This value is reported as cubic rack units (U) per liter (L); (U/L). Normal ranges are 6-29 U/L. Any participant with a value of 2 times or higher of the upper end of this range (58 U/L or greater) will be withdrawn from the study per study stopping criteria. This value will be reported as: "Number of participants with normal ALT levels," "Number of participants with abnormal ALT values," and "Number of participants withdrawn from the study based on elevated ALT values."
Estimated glomerular filtration rate (eGFR) | Mean change in Screening eGFR value at 4 weeks.
  Glomerular filtration rate is estimated based on blood creatinine concentration per standard nephrology practice. This value is reported as milliliters/minute/1.73m2 (mL/min/1.73m2). An eGFR value is considered normal if it is 60 or greater mL/min/1.73m2, and abnormal if it is less than 60 mL/min/1.73m2. Results will be reported as normal (60 or greater mL/min/1.73m2) or abnormal (less than 60 mL/min/1.73m2). Participants will be withdrawn from the study if two consecutive readings of eGFR show a decrease in eGFR of 15 mL/min/1.73m2 or greater.
Estimated glomerular filtration rate (eGFR) | Mean change in Screening eGFR value at 8 weeks.
  Glomerular filtration rate is estimated based on blood creatinine concentration per standard nephrology practice. This value is reported as milliliters/minute/1.73m2 (mL/min/1.73m2). An eGFR value is considered normal if it is 60 or greater mL/min/1.73m2, and abnormal if it is less than 60 mL/min/1.73m2. Results will be reported as normal (60 or greater mL/min/1.73m2) or abnormal (less than 60 mL/min/1.73m2). Participants will be withdrawn from the study if two consecutive readings of eGFR show a decrease in eGFR of 15 mL/min/1.73m2 or greater.
Estimated glomerular filtration rate (eGFR) | Mean change in 4 weeks eGFR value at 8 weeks.
  Glomerular filtration rate is estimated based on blood creatinine concentration per standard nephrology practice. This value is reported as milliliters/minute/1.73m2 (mL/min/1.73m2). An eGFR value is considered normal if it is 60 or greater mL/min/1.73m2, and abnormal if it is less than 60 mL/min/1.73m2. Results will be reported as normal (60 or greater mL/min/1.73m2) or abnormal (less than 60 mL/min/1.73m2). Participants will be withdrawn from the study if two consecutive readings of eGFR show a decrease in eGFR of 15 mL/min/1.73m2 or greater.
International normalized ratio | Mean change in Screening INR value at 4 weeks.
  Prothrombin time (PT) measures the ability of the blood to form blood clots through hemostasis. Partial thromboplastin time (PTT) also assess the ability to form blood clots through hemostasis, as well as amount and functions of proteins that initiate the clotting process (coagulation factors). PT and PTT will be combined to calculate the International Normalized Ratio (INR). INR is a calculation based on PT and PTT that measures the ability to form blood clots. INR values are dimensionless and will be reported numerically. A value less than 2.0 is considered normal. Any values of 2.0 or greater are considered abnormal and will result in exclusion from the study. If 25% or more of the study participants have INR values of 2.0 or greater at any point during the study period, the study will end and all participants will be withdrawn. Reported as numerical values of INR, percent of participants withdrawn from the study based on INR values of 2.0 or greater, and study stopping criteria.
International normalized ratio | Mean change in Screening INR value at 8 weeks.
  Prothrombin time (PT) measures the ability of the blood to form blood clots through hemostasis. Partial thromboplastin time (PTT) also assess the ability to form blood clots through hemostasis, as well as amount and functions of proteins that initiate the clotting process (coagulation factors). PT and PTT will be combined to calculate the International Normalized Ratio (INR). INR is a calculation based on PT and PTT that measures the ability to form blood clots. INR values are dimensionless and will be reported numerically. A value less than 2.0 is considered normal. Any values of 2.0 or greater are considered abnormal and will result in exclusion from the study. If 25% or more of the study participants have INR values of 2.0 or greater at any point during the study period, the study will end and all participants will be withdrawn. Reported as numerical values of INR, percent of participants withdrawn from the study based on INR values of 2.0 or greater, and study stopping criteria.
International normalized ratio | Mean change in 4 weeks INR value at 8 weeks.
  Prothrombin time (PT) measures the ability of the blood to form blood clots through hemostasis. Partial thromboplastin time (PTT) also assess the ability to form blood clots through hemostasis, as well as amount and functions of proteins that initiate the clotting process (coagulation factors). PT and PTT will be combined to calculate the International Normalized Ratio (INR). INR is a calculation based on PT and PTT that measures the ability to form blood clots. INR values are dimensionless and will be reported numerically. A value less than 2.0 is considered normal. Any values of 2.0 or greater are considered abnormal and will result in exclusion from the study. If 25% or more of the study participants have INR values of 2.0 or greater at any point during the study period, the study will end and all participants will be withdrawn. Reported as numerical values of INR, percent of participants withdrawn from the study based on INR values of 2.0 or greater, and study stopping criteria.
Systolic Blood pressure | Mean change from Baseline systolic blood pressure at 4 weeks.
  Blood pressure is used to assess hemodynamic stability by measuring the pressure of circulating blood on the walls of blood vessels. Systolic pressure will be assessed during the study period. Reported as: hypotension (less than 90 mmHg), normal blood pressure (90-139 mmHg), or hypertension (140 or greater mmHg). 2 consecutive readings of hypotension or hypertension will results in withdrawal from the study. Readings of systolic blood pressure from participants who complete the study will be reported in a table showing both systolic and diastolic readings at each time point assessed (Baseline and 4 weeks).
Systolic Blood pressure | Mean change from Baseline systolic blood pressure at 8 weeks.
  Blood pressure is used to assess hemodynamic stability by measuring the pressure of circulating blood on the walls of blood vessels. Systolic pressure will be assessed during the study period. Reported as: hypotension (less than 90 mmHg), normal blood pressure (90-139 mmHg), or hypertension (140 or greater mmHg). 2 consecutive readings of hypotension or hypertension will results in withdrawal from the study. Readings of systolic blood pressure from participants who complete the study will be reported in a table showing both systolic and diastolic readings at each time point assessed (Baseline and 8 weeks).
Systolic Blood pressure | Mean change from 4 weeks systolic blood pressure at 8 weeks.
  Blood pressure is used to assess hemodynamic stability by measuring the pressure of circulating blood on the walls of blood vessels. Systolic pressure will be assessed during the study period. Reported as: hypotension (less than 90 mmHg), normal blood pressure (90-139 mmHg), or hypertension (140 or greater mmHg). 2 consecutive readings of hypotension or hypertension will results in withdrawal from the study. Readings of systolic blood pressure from participants who complete the study will be reported in a table showing both systolic and diastolic readings at each time point assessed (4 weeks and 8 weeks).
Diastolic Blood pressure | Mean change from Baseline diastolic blood pressure at 4 weeks.
  Blood pressure is used to assess hemodynamic stability by measuring the pressure of circulating blood on the walls of blood vessels. Diastolic pressure will be assessed during the study period. Reported as: hypotension (less than 60 mmHg), normal blood pressure (60-89 mmHg), or hypertension (90 or greater mmHg). 2 consecutive readings of hypotension or hypertension will results in withdrawal from the study. Readings of blood pressure from participants who complete the study will be reported in a table showing both systolic and diastolic readings at each time point assessed (Baseline and 4 weeks).
Diastolic Blood pressure | Mean change from Baseline diastolic blood pressure at 8 weeks.
  Blood pressure is used to assess hemodynamic stability by measuring the pressure of circulating blood on the walls of blood vessels. Diastolic pressure will be assessed during the study period. Reported as: hypotension (less than 60 mmHg), normal blood pressure (60-89 mmHg), or hypertension (90 or greater mmHg). 2 consecutive readings of hypotension or hypertension will results in withdrawal from the study. Readings of blood pressure from participants who complete the study will be reported in a table showing both systolic and diastolic readings at each time point assessed (Baseline and 8 weeks).
Diastolic Blood pressure | Mean change from 4 weeks diastolic blood pressure at 8 weeks.
  Blood pressure is used to assess hemodynamic stability by measuring the pressure of circulating blood on the walls of blood vessels. Diastolic pressure will be assessed during the study period. Reported as: hypotension (less than 60 mmHg), normal blood pressure (60-89 mmHg), or hypertension (90 or greater mmHg). 2 consecutive readings of hypotension or hypertension will results in withdrawal from the study. Readings of blood pressure from participants who complete the study will be reported in a table showing both systolic and diastolic readings at each time point assessed (4 weeks and 8 weeks).

SECONDARY OUTCOMES:
Anxiety Subscore Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | Mean change in Baseline Anxiety Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) measures is a survey designed to measure self-reported physical, mental, and social health and wellbeing. This survey consists of 7 subscale scores, including: symptom-oriented subscores (anxiety, depression, fatigue, pain interference, and sleep disturbance) and function-oriented domains (physical functioning and social role). The anxiety subscale score ranges from 4-20, with a higher score indicating higher anxiety and a lower score indicating lower anxiety. Reported as a subscale.
Depression Subscore of the Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | Mean change in Baseline Depression Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) measures is a survey designed to measure self-reported physical, mental, and social health and wellbeing. This survey consists of 7 subscale scores, including: symptom-oriented subscores (anxiety, depression, fatigue, pain interference, and sleep disturbance) and function-oriented domains (physical functioning and social role). The depression subscale score ranges from 4-20, with a higher score indicating more depression and a lower score indicating less depression. Reported as a subscale.
Fatigue Subscore of the Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | Mean change in Baseline Fatigue Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) measures is a survey designed to measure self-reported physical, mental, and social health and wellbeing. This survey consists of 7 subscale scores, including: symptom-oriented subscores (anxiety, depression, fatigue, pain interference, and sleep disturbance) and function-oriented domains (physical functioning and social role). The fatigue subscale score ranges from 4-20, with a higher score indicating more fatigue and a lower score indicating less fatigue. Reported as a subscale.
Pain Interference Subscore of the Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | Mean change in Baseline Pain Interference Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) measures is a survey designed to measure self-reported physical, mental, and social health and wellbeing. This survey consists of 7 subscale scores, including: symptom-oriented subscores (anxiety, depression, fatigue, pain interference, and sleep disturbance) and function-oriented domains (physical functioning and social role). The pain interference subscale score ranges from 4-20, with a higher score indicating more pain interference and a lower score indicating less pain interference. Reported as a subscale.
Sleep Disturbance Subscore of the Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | Mean change in Baseline Sleep Disturbance Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) measures is a survey designed to measure self-reported physical, mental, and social health and wellbeing. This survey consists of 7 subscale scores, including: symptom-oriented subscores (anxiety, depression, fatigue, pain interference, and sleep disturbance) and function-oriented domains (physical functioning and social role). The sleep disturbance subscale score ranges from 4-20, with a higher score indicating more sleep disturbance and a lower score indicating less sleep disturbance. Reported as a subscale.
Physical Functioning Subscore of the Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | Mean change in Baseline Physical Functioning Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) measures is a survey designed to measure self-reported physical, mental, and social health and wellbeing. This survey consists of 7 subscale scores, including: symptom-oriented subscores (anxiety, depression, fatigue, pain interference, and sleep disturbance) and function-oriented domains (physical functioning and social role). The physical functioning subscale score ranges from 4-20, with a higher score indicating more physical function and a lower score indicating less physical function. Reported as a subscale.
Social Role Subscore of the Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | Mean change in Baseline Social Role Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) measures is a survey designed to measure self-reported physical, mental, and social health and wellbeing. This survey consists of 7 subscale scores, including: symptom-oriented subscores (anxiety, depression, fatigue, pain interference, and sleep disturbance) and function-oriented domains (physical functioning and social role). The social role subscale score ranges from 4-20, with a higher score indicating more ability to participate in social roles and activities and a lower score indicating less ability to participate in social roles and activities. Reported as a subscale.
Visual Analog Scale (VAS) | Mean change in Baseline VAS Score and 4 weeks.
  The Visual Analog Scale (VAS) is a psychometric response scale used to measure the intensity of pain. Pain is a subjective measure and pain intensity is used to quantify how much a person believes they are in pain. This scale ranges from 0-10, with lower scores indicating less subjective pain and higher scores indicating more subjective pain. This will be reported as change in a numerical value.
Visual Analog Scale (VAS) | Mean change in Baseline VAS Score and 8 weeks.
  The Visual Analog Scale (VAS) is a psychometric response scale used to measure the intensity of pain. Pain is a subjective measure and pain intensity is used to quantify how much a person believes they are in pain. This scale ranges from 0-10, with lower scores indicating less subjective pain and higher scores indicating more subjective pain. This will be reported as change in a numerical value.
Visual Analog Scale (VAS) | Mean change in 4 weeks VAS Score and 8 weeks.
  The Visual Analog Scale (VAS) is a psychometric response scale used to measure the intensity of pain. Pain is a subjective measure and pain intensity is used to quantify how much a person believes they are in pain. This scale ranges from 0-10, with lower scores indicating less subjective pain and higher scores indicating more subjective pain. This will be reported as change in a numerical value.
Patient Reported Outcomes Measurement Information System (PROMIS) Sexual Function Measure | Mean change in Baseline PROMIS Sexual Function Score and 8 weeks.
  The Patient Reported Outcomes Measurement Information System (PROMIS) Sexual Function Measure measures sexual function and evaluation of sexual experiences over the past 30 days. It is a subjective measure with 10 questions. These include domains such as: interest in sexual activity, lubrication during sexual activity, physical comfort during sexual activity, physical pain during sexual activity, orgasm during sexual activity, and overall satisfaction with sexual activity. This measure is scored using the HealthMeasures Scoring Device, with higher scores indicating better sexual function and lower scores indicating worse sexual function.

OTHER OUTCOMES:
High sensitivity C-reactive protein (hs-CRP) | Mean change in Baseline hs-CRP and 8 weeks.
  hs-CRP measures tissue inflammation and injury. This measure is used in standard cardiac practices to assess risk of cardiovascular disease, inflammation, and injury. This value is reported as milligrams per liter (mg/L). A value of less than 3 mg/L indicates average risk of cardiovascular disease and inflammation and a value of 3 mg/L or greater indicates an increased risk of cardiovascular disease and inflammation. This will be reported as "Number of participants with normal risk of cardiovascular disease and inflammation," "Number of participants with higher risk of cardiovascular disease and inflammation," "Change in number of participants with higher risk of cardiovascular disease and inflammation to lower risk of cardiovascular disease and inflammation," and "Change in number of participants with normal risk of cardiovascular disease and inflammation to higher risk of cardiovascular disease and inflammation, reported as a percentage."
Prostaglandins | Mean change in Baseline prostaglandin levels and 8 weeks
  Prostaglandins are a group of hormone-like substances that act as a principal mediator of inflammation in diseases and in menstruation. Changes in the level of prostaglandins directly correlate with the amount of pain that may be subjectively experienced. The normal range of this value is 200-400 picograms per milliliter (pg/mL). This will be reported as: "Number of participants with normal prostaglandin levels," "Number of participants with elevated prostaglandin levels," "Number of participants with decreased prostaglandin values," "Number of participants whose prostaglandin levels decreased," and "Number of participants whose prostaglandin levels increased."

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, MPH, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Background] Osayande AS, Mehulic S. Diagnosis and initial management of dysmenorrhea. Am Fam Physician. 2014 Mar 1;89(5):341-6. PMID 24695505
- [Background] Zahradnik HP, Hanjalic-Beck A, Groth K. Nonsteroidal anti-inflammatory drugs and hormonal contraceptives for pain relief from dysmenorrhea: a review. Contraception. 2010 Mar;81(3):185-96. doi: 10.1016/j.contraception.2009.09.014. Epub 2009 Nov 6. PMID 20159173
- [Background] Halter F, Tarnawski AS, Schmassmann A, Peskar BM. Cyclooxygenase 2-implications on maintenance of gastric mucosal integrity and ulcer healing: controversial issues and perspectives. Gut. 2001 Sep;49(3):443-53. doi: 10.1136/gut.49.3.443. PMID 11511570
- [Background] Lee JH, Cheong J, Park YM, Choi YH. Down-regulation of cyclooxygenase-2 and telomerase activity by beta-lapachone in human prostate carcinoma cells. Pharmacol Res. 2005 Jun;51(6):553-60. doi: 10.1016/j.phrs.2005.02.004. PMID 15829436
- [Background] Twardowschy A, Freitas CS, Baggio CH, Mayer B, dos Santos AC, Pizzolatti MG, Zacarias AA, dos Santos EP, Otuki MF, Marques MC. Antiulcerogenic activity of bark extract of Tabebuia avellanedae, Lorentz ex Griseb. J Ethnopharmacol. 2008 Aug 13;118(3):455-9. doi: 10.1016/j.jep.2008.05.013. Epub 2008 May 18. PMID 18579323
- [Background] Pereira IT, Burci LM, da Silva LM, Baggio CH, Heller M, Micke GA, Pizzolatti MG, Marques MC, Werner MF. Antiulcer effect of bark extract of Tabebuia avellanedae: activation of cell proliferation in gastric mucosa during the healing process. Phytother Res. 2013 Jul;27(7):1067-73. doi: 10.1002/ptr.4835. Epub 2012 Sep 12. PMID 22969019
- [Background] Giacomelli I, Scartoni D, Fiammetta M, Baki M, Zei G, Muntoni C, Cappelli S, Greto D, Scoccianti S, Livi L. Oral Lapacho-Based Medication: An Easy, Safe, and Feasible Support to Prevent and/or Reduce Oral Mucositis During Radiotherapy for Head and Neck Cancer. Nutr Cancer. 2015;67(8):1247-53. doi: 10.1080/01635581.2015.1082114. Epub 2015 Oct 9. PMID 26451712
- [Background] Lee MH, Choi HM, Hahm DH, Her E, Yang HI, Yoo MC, Kim KS. Analgesic and anti-inflammatory effects in animal models of an ethanolic extract of Taheebo, the inner bark of Tabebuia avellanedae. Mol Med Rep. 2012 Oct;6(4):791-6. doi: 10.3892/mmr.2012.989. Epub 2012 Jul 17. PMID 22825254
- [Background] de Miranda FG, Vilar JC, Alves IA, Cavalcanti SC, Antoniolli AR. Antinociceptive and antiedematogenic properties and acute toxicity of Tabebuia avellanedae Lor. ex Griseb. inner bark aqueous extract. BMC Pharmacol. 2001;1:6. doi: 10.1186/1471-2210-1-6. Epub 2001 Sep 13. PMID 11574048
- [Background] Lira AA, Sester EA, Carvalho AL, Strattmann RR, Albuquerque MM, Wanderley AG, Santana DP. Development of lapachol topical formulation: anti-inflammatory study of a selected formulation. AAPS PharmSciTech. 2008;9(1):163-8. doi: 10.1208/s12249-007-9002-z. Epub 2008 Jan 25. PMID 18446477
- [Background] de Almeida ER, da Silva Filho AA, dos Santos ER, Lopes CA. Antiinflammatory action of lapachol. J Ethnopharmacol. 1990 May;29(2):239-41. doi: 10.1016/0378-8741(90)90061-w. No abstract available. PMID 2374436